CLINICAL TRIAL: NCT05767190
Title: The MotivAir Study: a Randomized Controlled Trial of Motivational Interviewing-Based Intervention to Improve Adherence to CPAP in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: The MotivAir Study to Improve CPAP Adherence in OSAS Patients
Acronym: MotivAir
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03J101
Record Dates: First submitted 2022-05-12; First posted 2023-03-14 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Sleep Apnea, Obstructive; Motivational Interviewing
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MotivAir group (Experimental): Subjects in the MotivAir group will follow an intervention - lasting approximately 45 minutes - based on motivational interviewing principles and techniques delivered by a trained nurse.
  Interventions: Behavioral: Motivational interviewing
- Treatment as usual (No Intervention): Participants assigned to the control group will receive a usual pulmonary rehabilitation program for patients with OSAS receiving CPAP therapy, which is a standard technical training comprising information regarding the use, maintenance and safety measures of the device, plus a home inspection delivered by a technician who has the only task of doing maintenance to the machinery.

INTERVENTIONS:
Behavioral: Motivational interviewing — During the intervention, the trained-nurse will provide a motivational interviewing-based intervention consisting of one session divided into two parts: educational (the concepts of sleep apnea and the symptoms, and the CPAP treatment will be focused on) and training activity (using MI not directly advocate for behavioral change (i.e., use CPAP as prescribed), but asks key questions to help the patient explore conflicting feelings about the change, weighs the positive consequences and negatives of this change, and allows the patient to realize the discrepancy between current risk behavior (i.e. not using CPAP as directed) and the patient's self-identified goals. The intervention will be tailored on the patient's stage of change based on Prochaska and DiClemente transtheoretical model (1982), in fact, the nurse will use MI not only at the beginning of therapy but also in every contact with the patient throughout the treatment (subsequent follow-up visits, phone calls, etc.).
  Arms: MotivAir group

SUMMARY:
This study aims to evaluate the effectiveness of the MotivAir program an intervention based on Motivational Interviewing (MI) principles and techniques - in enhancing adherence to Continuous Positive Airway Pressure (CPAP) therapy among patients with Obstructive Sleep Apnea Syndrome (OSAS).

Methods. A multicenter randomized controlled trial (RCT) design with random allocation at the level of the individual will be conducted to compare the impact of the experimental program (usual care plus MI) with a control group receiving usual care only in improving selected clinical and psychological parameters in the patients.

A minimum sample of 80 participants (40 patients per group) will be recruited in each center according to the inclusion criteria. After the initial screening, participants will be randomly assigned to either the experimental group or the control condition. The program will last 180 days and will be delivered by a trained nurse. The impact of the MotivAir program on selected primary (adherence to CPAP in terms of average hours of usage per night and the Apnea-Hypopnea Index, AHI) and secondary (motivation, perceived competence, quality of life, sleepiness, as well as the emotional state, daily life activities, and quality of the social relationships of the person) outcomes will be measured at baseline, and after 1-, 3-, and 6-month from CPAP initiation

DETAILED DESCRIPTION:
Socio-demographic (age, level of studies, presence of caregiver at home), psychological (motivation and perceived competence) clinical variables (somnolence and apnoea-hypopnea index), and variables concerning the time the patient spends from home to the care center and the confidence in using electronic applications will be used to classify patients' adherence to treatment as low, moderate or high, and to create a tailored motivational treatment plan for the subjects assigned to the experimental group. Patients showing low adherence will receive a more intensive care plan, than those recognized as highly compliant with CPAP use. The results are patients with the "a" profile (characterized by autonomy and mobility, predisposition to remote-controlled follow-up), patients with the "b" profile (need for more intensity in follow-up), or patients with the "c" profile (more difficulties to move around and require more intensive treatment). Profile "d" was applied to patients who were professional drivers, as they require specific interventions based on their occupation (see Rudilla et al., 2021a).

Participants assigned to the control group will receive a usual pulmonary rehabilitation program for patients with OSAS receiving CPAP therapy, which is a standard technical training comprising information regarding the use, maintenance and safety measures of the device, plus a home inspection delivered by a technician who has the only task of doing maintenance to the machinery.

In addition, subjects in the MotivAir group will follow a telephone-based intervention - lasting approximately 45 minutes - based on MI principles and techniques delivered by a nurse. For the specific purpose of the study, the nurse will preliminarily receive 8 hours of MI training provided by two psychologists experts in the MI approach (authors GR and GP). During the training, the nurse will learn about the collaborative, evocative, and client-centered spirit of MI, and the characteristics that define each stage of change and will be instructed to apply the basic communication and listening skills of this approach (open-ended questions, affirmations, reflective listening, summarizing). Then she will learn to reinforce and elicit change talk, while also responding in ways that reduce counter-change talk and to roll with the patients' inner resistance to change by affirming the patients' autonomy and reflecting their resistant speech with empathy. Next, the issues of how and when to introduce the development of a change plan, and enhance the individuals' commitment to change will be addressed.

The treatment plan will be implemented based on each patient's level of adherence. To low adherence (score below 16 on the ESS and CEPCA questionnaires) a more intensive telephone-based assistance (day 1, 8, 16, 30, 90, 120, 180 from the end of the rehabilitation period) will follow. In the case of high adherence (score greater than or equal to 16 on the ESS and CEPCA questionnaires), phone encounters will be set on days 1, 8, 30, 90, and 180 after treatment termination.

At 1-, 3- and 6-month follow-up, adherence to the device will be assessed by automatedly recorded CPAP usage (hours/night) and AHI. Changes in the selected psychological variable will be also examined.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of OSAS confirmed by polysomnography;
* being recommended for treatment with CPAP;
* being naïve to this type of intervention

Exclusion Criteria:

* use of oxygen therapy > 2 l/min;
* history of severe cognitive disorders;
* history of COPD: FEV1/FVC (Tiffeneau Index) ≤ 60% with FEV1 ≤ 50%;
* dyspnea on exertion (Borg > 6);
* diagnosis of Long Covid or Covid-19 infection < 4 months;
* chronic heart failure (NYHA: Grade III and IV);
* unstable ischemic heart disease;
* inability to understand the consent to participate;
* patient refusal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline adherence to CPAP at 6 months | 6 months from CPAP initiation
  average hours of usage per night
Change from baseline Apnea-Hypopnea Index (AHI) at 6 months | 6 months from CPAP initiation
  severity of apnea-hypopnea

SECONDARY OUTCOMES:
Change from baseline Motivation to change at 6 months | 6 months from CPAP initiation
  the need for changes in your lifestyle to make it healthier with a single item
Change from baseline of Evaluation of Perceived Competence in Adherence to CPAP in OSAS at 3 and 6 months | 6 months from CPAP initiation
  self-efficacy in overcoming barriers associated with the use of the cpap
Change from Baseline of Visual Analogical Well-being Scale for apnea at 6 months | 6 months from CPAP initiation
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Castelnuovo, PhD, Principal Investigator — Istututo Auxologico Italiano
Locations (1):
- San Giuseppe Hospital, Istituto Auxologico Italiano IRCSS, Verbania, Italy

IPD SHARING:
Plan to Share IPD: No
Results of the study published in a repository and in an International Journal